CLINICAL TRIAL: NCT06265194
Title: A Randomized Controlled Trial of Eye Movement Desensitization and Reprocessing (EMDR) in the Treatment of Fibromyalgia
Brief Title: Effect of EMDR in the Treatment of Fibromyalgia
Acronym: EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Therapeutic Sciences, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZAT2024
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: EMDR; RCT; Depression; Pain
MeSH Terms: conditions — Fibromyalgia; Depression; Pain | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Eligible participants were randomized into two groups: one receiving TAU treatment (control group) and the other receiving both TAU and EMDR (experimental group).
Who Masked: Participant
Masking Description: Participants do not have the knowledge of group interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (TAU and EMDR) (Experimental): Intervention Group: Received TAU and EMDR Therapists delivering EMDR Therapy provided psychotherapeutic services to clients in the experimental group using the EMDR Fibromyalgia Treatment.
  Interventions: Behavioral: EMDR; Behavioral: TAU
- Control (TAU) (Active Comparator): Control Group: TAU Routine fibromyalgia treatments, referred to as Treatment as Usual (TAU) in this study, were initiated in the outpatient clinic conditions. TAU are treatments designed by rheumatologists in accordance with current rheumatology guidelines.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: EMDR — The fibromyalgia protocol applied to the patients in the study was developed specifically for fibromyalgia by Konuk, and colleagues (Konuk et al.). In addition to the article, the details of the protocol and the study sheet are presented supplementary. After a short introduction, the participants were informed about the protocol, their -consent was obtained for registration, and a visual, tactile and audio bilateral stimulus that will be used in the application was introduced.
  Arms: Intervention (TAU and EMDR)
Behavioral: TAU — Treatment as Usual (TAU): Routine fibromyalgia treatments, referred to as Treatment as Usual (TAU) in this study, were initiated in the outpatient clinic conditions. TAU are treatments designed by rheumatologists in accordance with current rheumatology guidelines.

SUMMARY:
The goal of this randomized-controlled study is to investigate the impact of EMDR therapy on fibromyalgia symptoms, depression, sleep quality, and traumatic stress in fibromyalgia patients.

The main questions it aims to answer are:

* Does EMDR become useful in relieving pain and complaints in fibromyalgia patients?
* Is specific EMDR Fibromyalgia Protocol effective of fibromyalgia patients?
* Does EMDR therapy decrease depression, sleep quality and traumatic stress symptoms of individuals with fibromyalgia?

DETAILED DESCRIPTION:
Background: In addition to pharmacological treatments, psychotherapeutic approaches are recommended for the treatment of fibromyalgia. There is a suggestion that Eye Movement Desensitization and Reprocessing (EMDR) therapy may be effective. This study aims to investigate the impact of EMDR therapy on fibromyalgia symptoms, depression, sleep quality, and traumatic stress in fibromyalgia patients through a Randomized Controlled Study (RCT).

Material and methods: The sample for this study comprises 79 individuals diagnosed with fibromyalgia. Participants were randomly assigned to two groups: the 'Treatment as Usual' (TAU) group and the TAU+EMDR group. Prior to the study and at six different time points (before starting the study, at the end of the 5th, 10th, and 15th sessions, 1 month later, and 3 months later), participants completed assessments, including the Fibromyalgia Impact Questionnaire (FIQ), Visual Analog Scale (VAS), Fibromyalgia ACR 2010 Diagnostic Criteria (Widespread Pain Index (WPI) and Symptom Severity Scale (SSS)), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI), and Trauma Symptom Checklist-40 (TSC-40).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of fibromyalgia,
2. Age between 18-65,
3. Compliance with routine medical fibromyalgia treatment,
4. Cognitive and technical competence to meet the working conditions,
5. Volunteering to participate in the study.

Exclusion Criteria:

1. Receiving any psychotherapy,
2. Presence of psychiatric disorders such as Schizophrenia or Bipolar Affective Disorder, c) No other physical and psychological targets apart from trauma needing to be addressed before fibromyalgia pain (e.g., suicide, domestic violence, etc.),

d) Presence of an organic cause that can cause pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 1-month and 3-month follow-up.
  Patients with fibromyalgia pain who underwent the EMDR fibromyalgia protocol will exhibit greater improvement compared to the control group. The scores are between 0-4, and more scores mean worse results for the relevant items.
Pittsburgh Sleep Quality Index (PSQI) | 1-month and 3-month follow-up.
  The experimental group will show a significant reduction in sleep difficulties, and this improvement will persist in one-month and three-month follow-ups. The scores are between 0-3, and more scores mean worse results for the relevant items.
Trauma Symptom Checklist-40 (TSC-40) | 1-month and 3-month follow-up.
  Traumatic stress symptoms in fibromyalgia patients from the experimental group will significantly decrease after undergoing the EMDR Fibromyalgia Protocol. The scores are between 0-3, and more scores mean worse results for the relevant items.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 1-month and 3-month follow-up.
  The EMDR Fibromyalgia Protocol used in the study is not designed for depression primarily, however, even in this case, the level of depression will be decreased in the experimental group. The scores are between 0-3, and more scores mean worse results for the relevant items.

REFERENCES:
- [Derived] Zat Ciftci Z, Delibas DH, Kaya T, Kulcu DG, Sari A, Nazlikul H, Coskun Topsakal I, Aydin YE, Kavakci O, Savran C, Konuk E. A randomized controlled trial of Eye Movement Desensitization and Reprocessing (EMDR) Therapy in the treatment of fibromyalgia. Front Psychiatry. 2024 May 21;15:1286118. doi: 10.3389/fpsyt.2024.1286118. eCollection 2024. PMID 38835548